CLINICAL TRIAL: NCT01530867
Title: Physician-Patient Communication Project
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Derjung Tarn, Assistant Professor, University of California, Los Angeles
Other Study IDs: R01AT005883-02 (NIH); R01AT005883-02 (NIH)
Record Dates: First submitted 2012-01-02; First posted 2012-02-10 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Dietary Supplements
Keywords: Dietary Supplements; Physician-patient communication; Qualitative study; Audio recorded office visits

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Over half of all Americans take dietary supplements (vitamins, minerals, herbal products) along with their prescription medications. With the economic downturn, dietary supplement sales have surged, perhaps as a result of people attempting to stave off or delay medical care. Supplements are generally thought to be harmless, but some can potentially interact with prescription medications, cause liver or kidney damage, and even adversely affect surgical outcomes. Those substituting dietary supplements for prescription medications also may suffer significant adverse consequences. The United States Food and Drug Administration and the Institute of Medicine recommend that patients considering dietary supplement use consult their providers. Unfortunately, patients fail to disclose dietary supplement use in up to two-thirds of outpatient office visits. To improve discussions, it is important to understand what prompts physicians and patients to communicate about dietary supplements.

The overall objectives of this application are to understand how, when and why physicians and patients communicate about dietary supplements, and to assess how patients respond to these discussions. An ethnically diverse group of patients and their physicians will be surveyed and their office visits will be audio recorded. Audio recordings of the visits will be used to assess the relationship of patient and physician attitudes and values, and the physician-patient relationship on dietary supplement discussions. A subset of these patients and physicians will be interviewed to explore how they made decisions to initiate or forgo discussions about supplements. They also will be asked questions concerning the necessity of and responsibility for initiating dietary supplement conversations. Patient responses and reactions to actual discussions also will be explored. Data from observed and reported interactions will be compared to provide a deeper understanding of factors related to disclosure. This project aims to provide a broad understanding of the content of physician-patient discussions about dietary supplements, and to describe how and why physician and patient attitudes and opinions affect these discussions. Identification of mutable factors can result in interventions to increase communication about dietary supplements, help maintain patient safety, and promote appropriate use of supplements concurrent with prescription medications.

DETAILED DESCRIPTION:
Sixty one primary care and integrative or complementary and alternative medicine physicians will be recruited for the study. For each participating physician, ten patients will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish-speaking
* Aged 18 and older

Exclusion Criteria:

* Does not speak English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care physicians Integrative medicine / complementary and alternative medicine physicians Patients aged 18 and older of physicians participating in the study
Sampling Method: Non-Probability Sample
Enrollment: 456 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
patients disclosing dietary supplement use | Disclosure will be measured at a single time point - on the day the patient's office visit is audio recorded. A subset of patients will be selected for a semi-structured interview up to 1 week after the visit.
  Number of patients who disclosed dietary supplement use during audio recorded office visit

CONTACTS AND LOCATIONS:
Overall Officials: Derjung M Tarn, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (5):
- United States (5):
  - Kaiser Permanente LAMC, Los Angeles, California
  - Center for East-West Medicine, Los Angeles, California
  - LA Net Practice Based Research Network, Los Angeles, California
  - Community-based provider offices, Los Angeles, California
  - University of California, Los Angeles, Santa Monica, California